CLINICAL TRIAL: NCT06231979
Title: Effects of Adding Dexmedetomidine to Bupivacaine for Bilateral Erector Spinae Block in Lumbar Fusion Surgeries
Brief Title: Adding Dexmedetomidine to Bupivacaine for Bilateral Erector Spinae Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Hassan Refaat AL-Quossi, assistent lecture, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Erector Spinae Block
Record Dates: First submitted 2023-12-24; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Erector Spinae Block; Lumbar Fusion Surgeries; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will receive US-guided ESPB with 18 mL of bupivacaine 0.25 % and 1 μg/kg DEX diluted with saline to reach total volume 20 mL per side.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain
- Bupivacaine group (Experimental): Patients will receive US-guided ESPB with 18 mL of bupivacaine 0.25 % and 2 mL normal saline 0.9 % per side as control group.
  Interventions: Drug: Bupivacain; Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — 1 μg/kg Dexmedetomidine per side in erector spinae block
  Other Names: DEX
  Arms: Dexmedetomidine group
Drug: Bupivacain — 18 mL of bupivacaine 0.25 % per side in erector spinae block
  Other Names: Bup
Drug: Normal saline — 2 ml normal saline 0.9% per side in erector spinae block
  Other Names: Normal saline sodium chloride 0.9%
  Arms: Bupivacaine group

SUMMARY:
The aim of this study is to compare the analgesic effect of bilateral US-guided ESPB using bupivacaine alone versus bupivacaine and DEX in lumbar fusion surgeries.

DETAILED DESCRIPTION:
Surgical treatment of adult lumbar spinal disorders is associated with a substantial risk of perioperative complications. The improvement in management and the development of new techniques in anesthesia and surgical sciences have led to substantial reduction of complications related to lumbar spine surgeries.

Understanding these complications is important and valuable for both the patient and the surgeon. Nevertheless, complications represent undesirable consequences of lumbar spine surgery in adult patients.

Degenerative lumbar disease is one of the most common chronic diseases worldwide. The general incidence of lumbar stenosis accompanied by a significant deterioration in the quality of life reaches 5 % among patients aged < 50 years and approximately 10 - 15 % among elderly patients (50 - 70 years old) Moreover, lumbar stenosis appears to be one of the most common causes of decompression and fusion interventions in the lumbar spine in > 50 years old patients Lumbar surgeries refer to any type of surgical intervention involving any lumbar spine or lower back (between one or more of the L1 - S1 level), including operations for trauma and deformity. The complexity of procedures leads to an increase in comorbidities Major lumbar spine surgery causes severe postoperative pain, which typically persists for at least three days Risk factors most frequently associated with mortality include but are not limited to patients' age, sex, and comorbidity status Postoperative pain is one of the most troublesome pains for the surgical patients and is one of the causes of morbidity and prolonged hospital stay. Various studies have reported that maximal pain occurs in the first 4 postoperative hours and gradually declines by the third postoperative day .

Opiates and non-steroidal anti-inflammatory drugs have been routinely used across the world. Recent resurge of regional anesthetic techniques offer some advantages, especially reduced postoperative nausea and vomiting and less sedation .

Ultrasound (US)-guided erector spinae plane blockade (ESPB) was first developed by Forero in 2016 as an easy and safe way of managing thoracic neuropathic pain. Since that time, this block has gained in popularity and has been used to effectively provide analgesia for a variety of surgeries, including spine surgery .

Erector spinae plane blockade may also have a better safety profile when compared with neuraxial analgesia, perhaps because of direct visualization of the needle under ultrasonography guidance and the ease of placement, although this has not been decisively proven One disadvantage of this block is the short duration of action after a single injection Dexmedetomidine (DEX), is a highly selective and potent central alpha-2 adrenergic receptor agonist. Administration of this adjuvant in miscellaneous methods has received considerable attention in recent years Due to its analgesic and sedative effects, besides the lack of any respiratory-sparing effects, administration of this adjuvant is effective in reducing the need for opioids in the perioperative period and may even result in cooperative sedation.

The neuraxial administration of dexmedetomidine has nociceptive effects on somatic and visceral pains. It also reduces postoperative pain and prolongs analgesia.

Local anesthetic combined with DEX has been reported to prolong analgesia following several blocks. However, it is presently unclear whether adjuncts such as DEX will significantly prolong the duration of ESPB in lumbar fusion surgery.

Oxidative stress is a condition caused by an imbalance between the production and accumulation of reactive oxygen species (ROS) and the body's ability to detoxify these products.

An excess of ROS causes damage to all cellular components. The process of oxidative stress causes the peroxidation of lipids and proteins, the formation of lipid peroxides, DNA fragmentation, and the development of cell death.

ROS activity is usually assessed indirectly by measuring stable products derived from the interaction of these radicals with cellular components. The most-studied cellular antioxidants are superoxide dismutase (SOD) , glutathione peroxidase 1 (GPX1) and human malondialdehyde (MDA).

These enzymes provide the first line of defense against tissue damage caused by ROS. As part of the antioxidant pathway, SOD accelerates the conversion of superoxide to H2O2, while catalase and GPX convert H2O2 to water. SOD and GPX can be measured in serum or plasma to establish the levels of oxidative stress and antioxidant capacity of the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* age between 18-65 years
* American Society of Anesthesiologists (ASA) physical status I-II**
* scheduled for lumbar spine fusion surgeries ( 2 or 3 level lumbar fusion with or without decompression ) under general anesthesia .

Exclusion Criteria:

* Patient refusal.
* Patient with chronic use of opioid analgesia.
* Uncooperative patients with communication difficulties, which might prevent a reliable postoperative assessment.
* Contraindication to regional anesthesia (bleeding disorder, use of any anticoagulants, local infection).

Known allergy to local anesthetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
the cummulative opioid consumption during first 48 h postoperatively. | 48 hours postoperatively.

SECONDARY OUTCOMES:
Change in stress marker Super Oxide Dismutase (SOD) . | 24 hours postoperative.
  Change in stress marker Super Oxide Dismutase (SOD) level in serum after centrifugation between preoperative at time of cannulation and 24h. Postoperative.
Postoperative pain score using Visual Analogue Scale (VAS). | immediately postoperative

OTHER OUTCOMES:
Change in stress marker Glutathione peroxidase 1 | 24 hours postoperative.
  Change in stress marker Glutathione peroxidase 1 level in serum after centrifugation between preoperative at time of cannulation and 24h. Postoperative.

REFERENCES:
- [Background] Kalff R, Ewald C, Waschke A, Gobisch L, Hopf C. Degenerative lumbar spinal stenosis in older people: current treatment options. Dtsch Arztebl Int. 2013 Sep;110(37):613-23; quiz 624. doi: 10.3238/arztebl.2013.0613. Epub 2013 Sep 13. PMID 24078855
- [Background] Liu C, Guo C, Meng F, Zhu Z, Xia W, Liu H. Perioperative risk factors related to complications of lumbar spine fusion surgery in elderly patients. BMC Musculoskelet Disord. 2023 Jul 14;24(1):573. doi: 10.1186/s12891-023-06689-z. PMID 37452304
- [Background] Dhillon KS. Spinal Fusion for Chronic Low Back Pain: A 'Magic Bullet' or Wishful Thinking? Malays Orthop J. 2016 Mar;10(1):61-68. PMID 28435551
- [Background] Proietti L, Scaramuzzo L, Schiro' GR, Sessa S, Logroscino CA. Complications in lumbar spine surgery: A retrospective analysis. Indian J Orthop. 2013 Jul;47(4):340-5. doi: 10.4103/0019-5413.114909. PMID 23960276
- [Background] El-Sadawy Ali Eid M, Ibrahim Mohamed Hashesh M and Ahmed El-Badawy Mohamed M. Comparative Study Between Bupivacaine Alone Versus Bupivacaine With Fentanyl, And Bupivacaine With Dexamethasone In Ultrasound Guided Erector Spinae Plane Block For Postoperative Pain Relief In Patients Undergoing Lumber Spine Surgeries. Al-Azhar Medical Journal. 2022;51(1):507-18.
- [Background] Poorman GW, Moon JY, Wang C, Horn SR, Beaubrun BM, Bono OJ, Francis AM, Jalai CM, Passias PG. Rates of Mortality in Lumbar Spine Surgery and Factors Associated With Its Occurrence Over a 10-Year Period: A Study of 803,949 Patients in the Nationwide Inpatient Sample. Int J Spine Surg. 2018 Oct 15;12(5):617-623. doi: 10.14444/5076. eCollection 2018 Oct. PMID 30364742
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Huang J, Liu JC. Ultrasound-guided erector spinae plane block for postoperative analgesia: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Apr 14;20(1):83. doi: 10.1186/s12871-020-00999-8. PMID 32290814
- [Background] Abdelbadie M. Analgesic efficacy of the erector spinae plane block using bupivacaine vs. bupivacaine/magnesium sulphate in patients undergoing lumbar spine surgery: a randomized, double-blinded comparative study. Anaesthesia, Pain & Intensive Care. 2022;26(4):439-44.
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Coviello A, Vargas M, Castellano G, Maresca A, Servillo G. Ultrasound-guided Erector Spinae Plane Block (US-ESPB)-Anesthetic block: Case report. Clin Case Rep. 2020 Sep 10;8(12):2885-2888. doi: 10.1002/ccr3.3253. eCollection 2020 Dec. PMID 33363844
- [Background] Stondell C, Roberto R. Erector Spinae Plane Blocks With Liposomal Bupivacaine for Pediatric Scoliosis Surgery. J Am Acad Orthop Surg Glob Res Rev. 2022 Jan 21;6(1):e21.00272. doi: 10.5435/JAAOSGlobal-D-21-00272. PMID 35061632
- [Background] Bhushan S, Huang X, Su X, Luo L, Xiao Z. Ultrasound-guided erector spinae plane block for postoperative analgesia in patients after liver surgery: A systematic review and meta-analysis on randomized comparative studies. Int J Surg. 2022 Jul;103:106689. doi: 10.1016/j.ijsu.2022.106689. Epub 2022 Jun 1. PMID 35662584
- [Background] Schnabel A, Reichl SU, Weibel S, Kranke P, Zahn PK, Pogatzki-Zahn EM, Meyer-Friessem CH. Efficacy and safety of dexmedetomidine in peripheral nerve blocks: A meta-analysis and trial sequential analysis. Eur J Anaesthesiol. 2018 Oct;35(10):745-758. doi: 10.1097/EJA.0000000000000870. PMID 30095549
- [Background] Kaye AD, Chernobylsky DJ, Thakur P, Siddaiah H, Kaye RJ, Eng LK, Harbell MW, Lajaunie J, Cornett EM. Dexmedetomidine in Enhanced Recovery After Surgery (ERAS) Protocols for Postoperative Pain. Curr Pain Headache Rep. 2020 Apr 2;24(5):21. doi: 10.1007/s11916-020-00853-z. PMID 32240402
- [Background] Gousheh M, Akhondzadeh R, Rashidi M, Olapour A, Moftakhar F. Comparison of Dexmedetomidine and Morphine as Adjuvants to Bupivacaine for Epidural Anesthesia in Leg Fracture Surgery: A Randomized Clinical Trial. Anesth Pain Med. 2019 Aug 27;9(4):e91480. doi: 10.5812/aapm.91480. eCollection 2019 Aug. PMID 31803587
- [Background] Gao X, Zhao T, Xu G, Ren C, Liu G, Du K. The Efficacy and Safety of Ultrasound-Guided, Bi-Level, Erector Spinae Plane Block With Different Doses of Dexmedetomidine for Patients Undergoing Video-Assisted Thoracic Surgery: A Randomized Controlled Trial. Front Med (Lausanne). 2021 Nov 25;8:577885. doi: 10.3389/fmed.2021.577885. eCollection 2021. PMID 34901039
- [Background] Pizzino G, Irrera N, Cucinotta M, Pallio G, Mannino F, Arcoraci V, Squadrito F, Altavilla D, Bitto A. Oxidative Stress: Harms and Benefits for Human Health. Oxid Med Cell Longev. 2017;2017:8416763. doi: 10.1155/2017/8416763. Epub 2017 Jul 27. PMID 28819546
- [Background] Su LJ, Zhang JH, Gomez H, Murugan R, Hong X, Xu D, Jiang F, Peng ZY. Reactive Oxygen Species-Induced Lipid Peroxidation in Apoptosis, Autophagy, and Ferroptosis. Oxid Med Cell Longev. 2019 Oct 13;2019:5080843. doi: 10.1155/2019/5080843. eCollection 2019. PMID 31737171
- [Background] Savic Vujovic K, Zivkovic A, Dozic I, Cirkovic A, Medic B, Srebro D, Vuckovic S, Milovanovic J, Jotic A. Oxidative Stress and Inflammation Biomarkers in Postoperative Pain Modulation in Surgically Treated Patients with Laryngeal Cancer-Pilot Study. Cells. 2023 May 14;12(10):1391. doi: 10.3390/cells12101391. PMID 37408225
- [Background] Bhattacharyya A, Chattopadhyay R, Mitra S, Crowe SE. Oxidative stress: an essential factor in the pathogenesis of gastrointestinal mucosal diseases. Physiol Rev. 2014 Apr;94(2):329-54. doi: 10.1152/physrev.00040.2012. PMID 24692350